CLINICAL TRIAL: NCT02175706
Title: DUrable Polymer-based STent CHallenge of Promus ElemEnt Versus ReSolute Integrity (DUTCH PEERS): Randomized Multicenter Trial in All-Comers Population Treated Within Eastern NeThErlands-2 (TWENTE-2).
Brief Title: DUrable Polymer-based STent CHallenge of Promus ElemEnt Versus ReSolute Integrity
Acronym: DUTCHPEERS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Thorax Centrum Twente (Other)
Responsible Party: Principal Investigator, Clemens von Birgelen, Professor, Thorax Centrum Twente
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1.6
Record Dates: First submitted 2013-11-27; First posted 2014-06-26 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Coronary Artery Disease; Angina Pectoris; Unstable Angina Pectoris; Acute Coronary Syndrome; Coronary Stenosis; Coronary Restenosis
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Angina, Unstable; Acute Coronary Syndrome; Coronary Stenosis; Coronary Restenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resolute Integrity® (Active Comparator): The coating of Resolute Integrity consists of zotarolimus as antiproliferative agent and the BioLinx® polymer system. This polymer system consists of a blend of three different polymers: (1) the hydrophobic C10 polymer, which aids in the control of drug release; (2) the hydrophilic C19 polymer, which supports biocompatibility; and (3) polyvinyl pyrro-lidinone, which increases the initial drug burst and enhances the elution rate.
  Interventions: Device: Resolute Integrity®
- Promus Element® (Active Comparator): Promus Element utilizes everolimus, which has been shown to reduce tissue proliferation in the coronary vessels following stent implantation.
  Promus Element is composed of the Element platform, a thin fluoropolymer coating, and Everolimus.
  Interventions: Device: Promus Element®

INTERVENTIONS:
Device: Resolute Integrity® — Biolinx-zotarolimus coating on a chobalt-cromium alloy stent platform that has a novel sinusoidal design.
  Other Names: Resolute Integrity® drug eluting stent
  Arms: Resolute Integrity®
Device: Promus Element® — fluoropolymer-everolimus coating on a novel stent platform made from a platinum-chromium alloy
  Other Names: Promus Element® drug eluting stent
  Arms: Promus Element®

SUMMARY:
Rationale:

The introduction of drug-eluting stents (DES) in the treatment of coronary artery disease has led to a significant reduction in morbidity but there are further demands on DES performance. Such demands are an optimized performance in very challenging coronary lesions; third generation DES were developed in an effort to further improve DES performance in such challenging lesions. Two CE-certified third generation DES (Resolute Integrity and Promus Element stents) are currently available; there are no data that indicate an advantage of one of these DES over the other.

Objective:

To investigate whether the clinical outcome is similar after implantation of the Promus Element versus the Resolute Integrity stent (non-inferiority hypothesis).

Study design:

Multicenter, prospective, randomized single-blinded study.

Study population:

Patients who require percutaneous coronary interventions (PCI) for the treatment of coronary stenoses with an indication for DES use, according to current guidelines and/or the operators clinical judgement. All clinical syndromes will be included.

Intervention:

In patients who are eligible for DES implantation, the type of DES implanted will be randomized (Resolute Integrity stent versus Promus Element stent). At the start of the study, both DES will also be used in routine clinical practice.

Main study endpoints:

The primary endpoint is the incidence of target vessel failure at one year follow-up. Target vessel failure (TVF) is a composite endpoint consisting of cardiac death, target vessel MI, or clinically driven target vessel revascularization. Further secondary clinical and angiographic endpoints will be investigated, defined in accordance with suggestions of the Academic Research Consortium (ARC). Of note, the angiographic assessment is based on clinically indicated projections only and results in no additional x-ray exposure. There is no routine angiographic follow-up. If angiographic data are available in patients who undergo symptom-driven re-catheterization, we will analyze these data to get insight into the mechanisms of potential DES restenosis.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients will receive the routine clinical treatment. As a consequence, the risks of this trial do not exceed the risks of any routine PCI procedure.

DETAILED DESCRIPTION:
1. OBJECTIVES

   Primary research questions To investigate whether the outcome after the randomized implantation of the Resolute Integrity versus Promus Element drug-eluting stent are similar, as assessed in a non-inferiority setting by comparing target-vessel failure (TVF) of both stents at one year follow-up post stent implantation. In brief, we want to compare for both drug-eluting stents the combined endpoint of (1) cardiac death, (2) myocardial infarction that can be related to the target vessel or cannot be related to another vessel, and (3) clinically indicated revascularization related to the target-vessel. Based on the results of the RESOLUTE all-comers trial (the study stents in the RESOLUTE all comers trial used the same coatings and drugs used in the current trial but on different bare metal stent platforms), non-inferiority of Resolute Integrity and Promus Element is expected. This is not tested in a controlled randomized trial yet.

   Secondary research questions Effectivity, safety, clinical short- and long-term outcome, and the acute angiographic results of the implantation of two third-generation drug-eluting stents will be compared in a "real world", all-comers scenario. Angiographic comparison will be based on the routine coronary angiography runs recorded during diagnostic coronary angiography and PCI procedures. No additional mandatory angiographic studies after the index PCI are required.
2. STUDY DESIGN

   The DUTCH PEERS Study is a multi-center prospective single-blinded randomized study. Randomization will involve the type of DES used in study population. Patients will be blinded to the type DES they will receive. The general practitioner of the patient will be requested not to disclose this information to the patient. Analysts who perform the data analyses will be blinded to the type DES used as well.
3. STUDY POPULATION 3.1 Population (base) All patients who fulfil the inclusion criteria and undergo PCI with potential DES implantation will be asked to participate in the DUTCH PEERS, unless they meet one or more of the exclusion criteria.

Patients will receive a drug-eluting stent according to the guidelines (Guidelines NVVC/ESC) and/or the clinical decision of the interventional cardiologist.

3.2 Inclusion criteria

* Minimum age of 18 years
* Coronary artery disease and lesion(s) eligable for treatment with drug eluting stents according to clinical guidelines and/or the operators' judgement
* Patient is willing and able to cooperate with study procedures and required follow-up visits; and patient has been informed and agrees on the participation by signing an EC approved written informed consent.

3.3 Exclusion criteria

* Participation in another randomized drug or device study before reaching primary endpoint
* Planned surgery within 6 months of PCI unless dual antiplatelet therapy is maintained throughout the peri-surgical period
* intolerance to a P2Y12 receptor antagonist that results in the patient's inability to adhere to dual-antiplatelet therapy, or intolerance to aspirin, heparin, or components of the two DES examined.
* Known pregnancy
* Life expectancy of less than 1 year

4.1 Randomisation, blinding and treatment allocation Patients will be randomised by a computer program (block stratified randomization V5.0 by S. Piantadosi). The randomisation will be done in blocks of 8 and 4 in random order. No stratification will be employed. The study will be single blinded because the physician will know which stent is implanted. The patient will not know. Every attempt will be made to do all outcome assessments blinded. The analyst performing QCA and IVUS analysis will be blinded to the type of DES used.

Demographics and Medical Data

At baseline the data are collected by the researchers, research nurses, and/or nurse practitioners. Demographic and medical data are also collected by reviewing the patient's medical chart:

* demographics including: date of birth, gender, family history of cardiovascular disease, smoking habits;
* medical history including: arterial hypertension, diabetes mellitus, hypercholesterolemia, previous myocardial infarction, previous revascularization by means of CABG / PCI, previous cerebrovascular accident (CVA) or transient ischemic attack (TIA), renal failure requiring haemodialysis;
* current medication;
* body-mass index, arterial blood pressure, heart frequency;
* indication for PCI;
* symptoms prior to PCI: angina pectoris (CCS class), dyspnea (NYHA class).

Blood samples Laboratory tests will be performed in the local laboratories of the participating centres as part of their clinical routine practice. In elective and primary PCI before and the day after the PCI procedure, blood tests will be performed (assessment of Hb, Kreatinine, CK, CK-MB, and Troponines). If patients suffer from persistent chest pain after PCI, additional controls of the cardiac markers will be performed on the day of PCI as part of the clinical routine. In case of symptoms suspicious of an acute coronary event in patients scheduled for elective PCI, the assessment of cardiac markers prior to PCI is considered as good clinical practice and should be performed.

PCI procedure Routine PCI will be performed according to routine medical practice in including centres with no deviation from routine protocols. No additional angiographic views will be required. Patients will receive one or more DES during PCI. The type of DES used during PCI will be randomized. Detailed technical information on PCI procedures are provided in the current European society of cardiology guidelines of PCI. [27] If clinically indicated, IVUS-guidance will be used during PCI.

Mixture of stents should be avoided and is only permitted if the operator is unable to insert the study stent, in which case crossover to another non-study stent is possible. Treatment of all coronary lesions should be aimed in one session, however staged procedures (defined as procedures planned at the time of the index procedure and performed within 6 weeks with the same type of study stent) will be permitted. In case of unplanned revascularization procedures requiring stent implantation, it is recommended that physicians use the same study stent.

Medical therapy Medical therapy does not differ from current routine medical treatment. In brief, patients who are not on oral aspirin therapy receive a loading dose of at least 300 mg prior to PCI. In elective PCI patients, clopidogrel therapy of 75 mg daily is started one week before the PCI. In urgent PCI, a loading dose of 600 mg clopidogrel is given as soon as possible, either before PCI or (at least) directly after the PCI is performed. In case prasugrel is used, patients will receive a loading dose of 60 mg of prasugrel followed by a daily dose of 10 mg for at least 12 months. Directly prior to PCI, an adequate dose of unfractionated heparin is administered i.v. or i.a. In general, an intracoronary bolus of nitrates will be administered prior to PCI. The use of glycoprotein IIb/IIIa inhibitors is left at the operators' discretion. Following the index PCI procedure, patients are generally maintained on aspirin >=80 mg daily during the entire trial (and preferably lifelong). In general, clopidogrel 75 mg daily is recommended and prescribed for a period of 12 months in addition to aspirin. If patients require oral anticoagulation therapy (e.g. for atrial fibrillation), aspirin >=80 mg daily is prescribed for one month after PCI and clopidogrel for 12 months. Further medical treatment is performed according to current medical guidelines, clinical standards, and the judgment of the referring physicians.

Follow-up data collection Follow-up data will be collected during routine visits to outpatient clinic and/or phone calls. If no data are available from outpatient clinic visits, the required data will be collected through a phone call. The phone call follow-up will be conducted through blinded members of the research team (nurse practicioners, cardioresearch personnel or research fellows). Through an outpatient clinic visit or a telephone call patients will be asked about recurrence of symptoms or new symptoms which can indicate the presence of restenosis. Patients will be also asked about possible revascularization or myocardial infarction during the follow-up period. In case of death, information will be obtained from the patient's medical chart, GP or cardiologist. Patients will be called after 1 month, 12 months and 24 months. The mode of data acquisition of the follow up (telephone or outpatient visit) will be registered.

In order to determine whether a myocardial infarction is related or unrelated to the target vessel, a Critical Events Committee consisting of two independent cardiologists will be asked to provide an independent conclusion about the location of an infarction on the electrocardiogram.

Adverse events, comprised by the primary endpoint, will be monitored by an independent external contract research organisation. In addition, we intend that secondary clinical endpoints of at least 10% of patients will be monitored, too.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years;
* Coronary artery disease and lesion(s) eligable for treatment with drug eluting stents according to clinical guidelines and/or the operators' judgement;
* Patient is willing and able to cooperate with study procedures and required follow-up visits; and patient has been informed and agrees on the participation by signing an EC approved written informed consent.

Exclusion Criteria:

* Participation in another randomized drug or device study before reaching primary endpoint;
* Planned surgery within 6 months of PCI unless dual antiplatelet therapy is maintained throughout the peri-surgical period;
* Intolerance to aspirin, clopidogrel or ticlopidin, heparin, or components of the two DES examined;
* Known pregnancy;
* Life expectancy of less than 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1811 (Actual)
Dates: Start 2010-11; Primary Completion 2013-05 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Target-vessel failure (TVF) | 1 year
  Components of the primary endpoint in hierarchical order:
  1. Cardiac death. All deaths are considered cardiac, unless an unequivocal non-cardiac cause can be established;
  2. Target vessel related MI that is Q-wave or non-Q-wave myocardial infarction that can be related to the target vessel or cannot be related to another vessel;
  3. Clinically driven repeated target vessel revascularization by means of CABG or PCI.

SECONDARY OUTCOMES:
Death at 1 and 2 year follow-up | 1 and 2 year
  Death distinguished into: cardiac, vascular, other causes, all-cause mortality
Myocardial infarction at 1 and 2 year follow-up | 1 and 2 year
  Myocardial infarction distinguished into Q-wave and non-Q-wave myocardial infarction
Revascularization at 1 and 2 year follow-up | 1 and 2 year
  Target-vessel revascularization distinguished into PCI or CABG
Stent thrombosis at 1 and 2 year follow-up | 1 and 2 year
  Stent thrombosis was distinguished into definite, probable and possible according to the Academic Research Consortium (ARC) definition.

OTHER OUTCOMES:
Longitudinal stent deformation | 1 year
  Identification of deformation of a stent in the longitudinal axis during coronary angiographic assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Clemens von Birgelen, MD,PhD,Prof, Principal Investigator — Thorax Centrum Twente
Locations (4):
- Netherlands (4):
  - Medisch Centrum Alkmaar, Alkmaar
  - Ziekenhuis Rijnstate, Arnhem
  - Scheper Ziekenhuis, Emmen
  - Medisch Spectrum Twente, Enschede

IPD SHARING:
Plan to Share IPD: Undecided